CLINICAL TRIAL: NCT01467505
Title: A 2-Part, Open Label Study of Telaprevir in Combination With Peginterferon Alfa-2a (Pegasys®) and Ribavirin (Copegus®) in Subjects Chronically Infected With Genotype 1 Hepatitis C Virus Following Liver Transplantation
Brief Title: An Open Label Study of the Effect of Telaprevir in Combination With Ribavirin and Peginterferon on HCV Infection in Stable Liver Transplant Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated early by the sponsor on 13 January 2014 due to a decision to modify the drug development plan.
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VX11-950-117
Record Dates: First submitted 2011-11-03; First posted 2011-11-08 (Estimated); Results first posted 2015-06-18 (Estimated); Last update posted 2015-06-18 (Estimated); Status verified 2015-06

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — telaprevir; Ribavirin; peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- T/PR + Immunosuppressant Regimen (Tacrolimus) (Experimental): Participants who were receiving tacrolimus (TAC) based immunosuppressant regimen at baseline, received telaprevir (T) 1125 milligram (mg) tablet twice daily for 12 weeks in combination with pegylated interferon alfa 2a (P) (Peg-IFN-alfa-2a) 180 microgram per week (mcg/week) subcutaneous injection and ribavirin (R) (RBV) tablet orally twice daily at a dose of 1000 milligram per day (mg/day) for subjects weighing less than (<) 75 kilogram (kg) and 1200 mg/day for subjects weighing greater than or equal to (>=) 75 kg, for 48 weeks. Participants continued their immunosuppressant regimen, as per standard practice and investigator discretion.
  Interventions: Drug: Telaprevir; Drug: Ribavirin; Drug: Pegylated Interferon Alfa-2a; Drug: Immunosuppressant Regimen
- T/PR + Immunosuppressant Regimen (Cyclosporine) (Experimental): Participants who were receiving cyclosporine (CsA) based immunosuppressant regimen at baseline, received telaprevir 1125 mg tablet twice daily for 12 weeks in combination with Peg-IFN-alfa-2a 180 mcg/week subcutaneous injection and RBV tablet orally twice daily at a dose of 1000 mg/day for subjects weighing <75 kg and 1200 mg/day for subjects weighing >=75 kg, for 48 weeks. Participants continued their immunosuppressant regimen, as per standard practice and investigator discretion.
  Interventions: Drug: Telaprevir; Drug: Ribavirin; Drug: Pegylated Interferon Alfa-2a; Drug: Immunosuppressant Regimen

INTERVENTIONS:
Drug: Telaprevir — Tablet
  Other Names: VX-950
Drug: Ribavirin — Tablet
  Other Names: Copegus®, RBV
Drug: Pegylated Interferon Alfa-2a — Subcutaneous Injection
  Other Names: Pegasys®, Peg-IFN-alfa-2a
Drug: Immunosuppressant Regimen — Cyclosporine (CsA) based immunosuppressant regimen or Tacrolimus (TAC) based immunosuppressant regimen, as per standard practice. Immunosuppressant regimen were not considered study drugs.

SUMMARY:
To assess efficacy of telaprevir, pegylated interferon alfa-2a (Peg-IFN-alfa-2a), and ribavirin (RBV) for hepatitis C virus (HCV) in a 48-week total treatment duration regimen following liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants between the ages of 18 and 65 years
* History of orthotopic liver transplantation less than 10 years before the Screening visit but no sooner than 6 months before Day 1
* Taking a stable immunosuppressant regimen based on either tacrolimus or cyclosporine without substantial dose changes over the past 3 months
* Naive to pegylated interferon/ribavirin treatment or experienced with pegylated interferon/ribavirin prior to transplantation with relapse, partial, or null response

Exclusion Criteria:

* Documented cirrhosis after liver transplantation
* Ascites or hepatic encephalopathy within 6 months before Screening
* Retransplantation for recurrent hepatitis C
* Treatment for hepatitis C post liver transplantation
* History within the past 3 months of: rejection within 3 months or greater than (>) 1 rejection within 12 months
* Current treatment with sirolimus or methylprednisolone. Low dose prednisone use (<5 milligram per day) is permitted
* History within 3 months of any bacterial infection requiring >1 week of intravenous antibiotics, cytomegalovirus viremia or cytomegalovirus infection with end-organ involvement, fungal disease (except cutaneous and mild oral thrush)
* History of post transplant lymphoproliferative disease
* Acceptable laboratory values at Screening as specified in the protocol
* Positive for human immunodeficiency virus 1/2 (HIV1/2) enzyme immunoassay (EIA) antibody screen or Hepatitis B deoxyribonucleic acid (DNA) or Hepatitis B surface antigen
* History of hepatocellular carcinoma with high risk of recurrence
* Any other cause of liver disease deemed clinically significant by the investigator in addition to hepatitis C
* Autoimmune-mediated disease
* History of acute pancreatitis within 5 years before the Screening visit
* Prior treatment with an hepatitis C virus (HCV) protease inhibitor

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2012-02; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Vertex Pharmaceuticals Incorporated
Locations (22):
- United States (20):
  - Alabama, Birmingham, Alabama
  - Arizona, Phoenix, Arizona
  - California, Los Angeles, California
  - Colorado, Denver, Colorado
  - Florida, Bradenton, Florida
  - Florida, Miami, Florida
  - Illinios, Evanston, Illinois
  - Indiana, Indianapolis, Indiana
  - Massachusetts, Burlington, Massachusetts
  - Michigan, Ann Arbor, Michigan
  - Michigan, Detroit, Michigan
  - Missouri, St Louis, Missouri
  - Nebraska, Omaha, Nebraska
  - New York, New York, New York
  - New York, Rochester, New York
  - North Carolina, Charlotte, North Carolina
  - Ohio, Cleveland, Ohio
  - Pennsylvania, Philadelphia, Pennsylvania
  - Texas, Dallas, Texas
  - Texas, Houston, Texas
- Canada (2):
  - Calgary, Alberta
  - Vancouver, British Columbia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study included Treatment-Naïve (no prior hepatitis C virus [HCV] therapy); Prior Relapser (prior treatment with pegylated interferon alfa/ribavirin [Peg-IFN/RBV] and experienced viral relapse); Prior Null/Partial Responder (prior treatment with Peg-IFN/RBV and had null/partial response); Uncategorized (could not tolerate treatment) participants.
Pre-assignment Details: Efficacy analyses were reported separately as per immunosuppressant regimen (reporting arms) and also separately as per prior response (in categories) (Treatment-Naive, Prior Relapser, Prior Null Responder, Prior Partial Responder, Uncategorized as well as for Total Participants), unless otherwise specified.
Period: Overall Study
Arm/Group | T/PR + Immunosuppressant Regimen (Tacrolimus) | T/PR + Immunosuppressant Regimen (Cyclosporine)
Started | 51 | 10
Completed | 18 | 7
Not Completed | 33 | 3
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 4 | 0
Not completed — Study Terminated by Sponsor | 28 | 3

BASELINE CHARACTERISTICS:
Population: Full analysis set included all participants who received at least 1 dose of study drug.
Groups:
- T/PR + Immunosuppressant Regimen (Tacrolimus): Participants who were receiving TAC based immunosuppressant regimen at baseline, received telaprevir 1125 mg tablet twice daily for 12 weeks in combination with Peg-IFN-alfa-2a 180 mcg/week subcutaneous injection and RBV tablet orally twice daily at a dose of 1000 mg/day for subjects weighing <75 kg and 1200 mg/day for subjects weighing >=75 kg, for 48 weeks. Participants continued their immunosuppressant regimen, as per standard practice and investigator discretion.
- T/PR + Immunosuppressant Regimen (Cyclosporine): Participants who were receiving CsA based immunosuppressant regimen at baseline, received telaprevir 1125 mg tablet twice daily for 12 weeks in combination with Peg-IFN-alfa-2a 180 mcg/week subcutaneous injection and RBV tablet orally twice daily at a dose of 1000 mg/day for subjects weighing <75 kg and 1200 mg/day for subjects weighing >=75 kg, for 48 weeks. Participants continued their immunosuppressant regimen, as per standard practice and investigator discretion.
- Total: Total of all reporting groups
Arm/Group | T/PR + Immunosuppressant Regimen (Tacrolimus) | T/PR + Immunosuppressant Regimen (Cyclosporine) | Total
Number analyzed (Participants) | 51 | 10 | 61
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.8 (4.08) | 59.5 (2.95) | 57.3 (4.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 0 | 12
  Male | 39 | 10 | 49

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Viral Response 12 Weeks After Last Planned Dose of Study Drug (SVR12)
Description: SVR12 was defined as an undetectable Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) Levels (<lower limit of quantification) at 12 weeks after last planned dose of study treatment. The plasma HCV RNA level was measured using Roche TaqMan HCV RNA assay. The lower limit of quantification was 25 international units per milliliter (IU/mL).
Time Frame: 12 weeks after last planned dose of study drug (up to Week 60)
Population: Safety Set included all participants who received at least 1 dose of study drug. Here, n = participants evaluable for specified category for each arm, respectively.
Measure: Number; unit: percentage of participants
Arm/Group | T/PR + Immunosuppressant Regimen (Tacrolimus) | T/PR + Immunosuppressant Regimen (Cyclosporine)
Number analyzed (Participants) | 51 | 10
percentage of participants
  Naive (n= 16, 2) | 75.0 | 50.0
  Prior Relapser (n= 10, 2) | 60.0 | 100.0
  Prior Null Responder (n=16, 4) | 37.5 | 50.0
  Prior Partial Responder (n= 3, 1) | 66.7 | 100.0
  Uncategorized (n= 6, 1) | 50.0 | 100.0
  Total (n= 51, 10) | 56.9 | 70.0

2. Secondary Outcome: Percentage of Participants With Sustained Viral Response 24 Weeks After Last Planned Dose of Study Drug (SVR24)
Description: SVR24 was defined as an undetectable HCV RNA Levels at 24 weeks after last planned dose of study treatment. The plasma HCV RNA level was measured using Roche TaqMan HCV RNA assay. The lower limit of quantification was 25 IU/mL.
Time Frame: 24 weeks after last planned dose of study drug (up to Week 72)
Population: Safety Set included all participants who received at least 1 dose of study drug. Here, number of participants analyzed = participants evaluable for this measure and n = participants evaluable for specified category for each arm, respectively.
Measure: Number; unit: percentage of participants
Arm/Group | T/PR + Immunosuppressant Regimen (Tacrolimus) | T/PR + Immunosuppressant Regimen (Cyclosporine)
Number analyzed (Participants) | 24 | 7
percentage of participants
  Naive (n= 5,1) | 60.0 | 0
  Prior Relapser (n= 4,1) | 25.0 | 0
  Prior Null Responder (n=10, 4) | 20.0 | 50.0
  Prior Partial Responder (n= 0, 1) | 0 | 100.0
  Uncategorized (n= 5, 0) | 20.0 | 0
  Total (n= 24, 7) | 29.2 | 42.9

3. Secondary Outcome: Percentage of Participants With Rapid Viral Response (RVR)
Description: The plasma HCV RNA level was measured using Roche TaqMan HCV RNA assay. The lower limit of quantification was 25 IU/mL and the lower limit of detection was 10 IU/mL. RVR was defined as undetectable HCV RNA 4 weeks after the start of study treatment.
Time Frame: Week 4
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | T/PR + Immunosuppressant Regimen (Tacrolimus) | T/PR + Immunosuppressant Regimen (Cyclosporine)
Number analyzed (Participants) | 51 | 10
percentage of participants
  Naive (n= 16, 2) | 68.8 | 0
  Prior Relapser (n= 10, 2) | 50.0 | 50.0
  Prior Null Responder (n=16, 4) | 43.8 | 25.0
  Prior Partial Responder (n= 3, 1) | 66.7 | 100.0
  Uncategorized (n= 6, 1) | 33.3 | 0
  Total (n= 51, 10) | 52.9 | 30.0

4. Secondary Outcome: Percentage of Participants With Extended Rapid Viral Response (eRVR)
Description: The plasma HCV RNA level was measured using Roche TaqMan HCV RNA assay. The lower limit of quantification was 25 IU/mL and the lower limit of detection was 10 IU/mL. eRVR was defined as undetectable HCV RNA at both 4 weeks and 12 weeks after the start of study treatment.
Time Frame: Week 4 and Week 12
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | T/PR + Immunosuppressant Regimen (Tacrolimus) | T/PR + Immunosuppressant Regimen (Cyclosporine)
Number analyzed (Participants) | 51 | 10
percentage of participants
  Naive (n= 16, 2) | 68.8 | 0
  Prior Relapser (n= 10, 2) | 50.0 | 50.0
  Prior Null Responder (n=16, 4) | 37.5 | 25.0
  Prior Partial Responder (n= 3, 1) | 66.7 | 100.0
  Uncategorized (n= 6, 1) | 33.3 | 0
  Total (n= 51, 10) | 51.0 | 30.0

5. Secondary Outcome: Percentage of Participants With On-Treatment Virologic Failure
Description: On-treatment virologic failure was defined as subjects who met futility or who completed the assigned treatment duration and had detectable HCV RNA at planned end of treatment (up to 48 weeks). Data for this outcome was not planned to be reported by prior response.
Time Frame: Baseline up to Week 48
Population: Safety Set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | T/PR + Immunosuppressant Regimen (Tacrolimus) | T/PR + Immunosuppressant Regimen (Cyclosporine)
Number analyzed (Participants) | 51 | 10
percentage of participants | 0 | 0

6. Secondary Outcome: Percentage of Participants With Viral Relapse
Time Frame: 48 weeks
Population: Due to early study termination as part of a decision to modify the drug development plan the data for this outcome measure was not collected, as planned.
Arm/Group | T/PR + Immunosuppressant Regimen (Tacrolimus) | T/PR + Immunosuppressant Regimen (Cyclosporine)
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Pharmacokinetics of Telaprevir, Peg-IFN, RBV , and Selected Immunosuppressant Medications (Tacrolimus and Cyclosporine)
Time Frame: 48 weeks
Population: as for outcome 6
Arm/Group | T/PR + Immunosuppressant Regimen (Tacrolimus) | T/PR + Immunosuppressant Regimen (Cyclosporine)
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Percentage of Participants Requiring Dose Titration of Immunosuppressant Medications
Time Frame: 48 weeks
Population: as for outcome 6
Arm/Group | T/PR + Immunosuppressant Regimen (Tacrolimus) | T/PR + Immunosuppressant Regimen (Cyclosporine)
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Percentage of Participants With Biopsy Confirmed and Treated Rejection
Time Frame: 48 weeks
Population: as for outcome 6
Arm/Group | T/PR + Immunosuppressant Regimen (Tacrolimus) | T/PR + Immunosuppressant Regimen (Cyclosporine)
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Percentage of Participants With Histological Evidence of Stabilization or Improvement in Inflammation Grade or Fibrosis Stage
Time Frame: 48 weeks
Population: as for outcome 6
Arm/Group | T/PR + Immunosuppressant Regimen (Tacrolimus) | T/PR + Immunosuppressant Regimen (Cyclosporine)
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Number of Participants With Telaprevir Resistant HCV Variant at Non-Structural Viral Protein 3-4A (NS3-4A) Region
Time Frame: 48 weeks
Population: as for outcome 6
Arm/Group | T/PR + Immunosuppressant Regimen (Tacrolimus) | T/PR + Immunosuppressant Regimen (Cyclosporine)
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Any adverse change from the participant's baseline (pre-treatment) condition, including any adverse experience, abnormal recording or clinical laboratory assessment value which occurs during the course of the study, whether it is considered related to the study drug or not. An adverse event includes any newly occurring event or previous condition that has increased in severity or frequency since the administration of study drug. SAE: medical event or condition, which falls into any of the following categories, regardless of its relationship to the study drug: death, life threatening adverse experience, in-patient hospitalization/prolongation of hospitalization, persistent/significant disability or incapacity, congenital anomaly/birth defect, important medical event. "Study drug" includes all investigational agents (including placebo, if applicable) administered during the course of the study.
Time Frame: Baseline up to Week 52
Population: Safety Set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | T/PR + Immunosuppressant Regimen (Tacrolimus) | T/PR + Immunosuppressant Regimen (Cyclosporine)
Number analyzed (Participants) | 51 | 10
participants
  AEs | 51 | 10
  SAEs | 11 | 3

13. Other Pre Specified Outcome: Percentage of Participants With Sustained Viral Response 4 Weeks After Last Planned Dose of Study Drug (SVR4)
Time Frame: 4 weeks after last planned dose of study drug (up to Week 52)
Population: as for outcome 6
Arm/Group | T/PR + Immunosuppressant Regimen (Tacrolimus) | T/PR + Immunosuppressant Regimen (Cyclosporine)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to Week 52
Description: Other Adverse Events section includes both Serious Adverse Events (SAEs) and Non-Serious Adverse Events (Non-SAEs) as Non-SAEs were not planned to be summarized separately for this study.
Arm/Group | T/PR + Immunosuppressant Regimen (Tacrolimus) | T/PR + Immunosuppressant Regimen (Cyclosporine)
Serious Adverse Events (participants affected / at risk) | 11/51 | 3/10
Other Adverse Events (participants affected / at risk) | 51/51 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | T/PR + Immunosuppressant Regimen (Tacrolimus) (N=51) | T/PR + Immunosuppressant Regimen (Cyclosporine) (N=10)
Nausea (Gastrointestinal disorders) | 4 | 0
Vomiting (Gastrointestinal disorders) | 4 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 2 | 0
Herpes zoster (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1
Pain (General disorders) | 1 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Irritability (Psychiatric disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | T/PR + Immunosuppressant Regimen (Tacrolimus) (N=51) | T/PR + Immunosuppressant Regimen (Cyclosporine) (N=10)
Nausea (Gastrointestinal disorders) | 29 | 4
Diarrhoea (Gastrointestinal disorders) | 24 | 3
Anorectal discomfort (Gastrointestinal disorders) | 14 | 3
Anal pruritus (Gastrointestinal disorders) | 7 | 4
Vomiting (Gastrointestinal disorders) | 9 | 2
Abdominal pain (Gastrointestinal disorders) | 8 | 0
Constipation (Gastrointestinal disorders) | 6 | 0
Dyspepsia (Gastrointestinal disorders) | 5 | 1
Dry mouth (Gastrointestinal disorders) | 4 | 1
Abdominal distension (Gastrointestinal disorders) | 2 | 2
Flatulence (Gastrointestinal disorders) | 3 | 1
Proctalgia (Gastrointestinal disorders) | 3 | 1
Abdominal discomfort (Gastrointestinal disorders) | 2 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 2
Abdominal pain lower (Gastrointestinal disorders) | 2 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 0
Glossitis (Gastrointestinal disorders) | 1 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 0
Abdominal hernia (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Abdominal tenderness (Gastrointestinal disorders) | 1 | 0
Bowel movement irregularity (Gastrointestinal disorders) | 1 | 0
Chapped lips (Gastrointestinal disorders) | 1 | 0
Cheilitis (Gastrointestinal disorders) | 1 | 0
Faeces discoloured (Gastrointestinal disorders) | 1 | 0
Faeces soft (Gastrointestinal disorders) | 1 | 0
Frequent bowel movements (Gastrointestinal disorders) | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 1 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 1
Haematochezia (Gastrointestinal disorders) | 1 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 0
Lip swelling (Gastrointestinal disorders) | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0
Mucous stools (Gastrointestinal disorders) | 1 | 0
Oral mucosal blistering (Gastrointestinal disorders) | 1 | 0
Palatal disorder (Gastrointestinal disorders) | 1 | 0
Perianal erythema (Gastrointestinal disorders) | 1 | 0
Retching (Gastrointestinal disorders) | 1 | 0
Swollen tongue (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 36 | 7
Influenza like illness (General disorders) | 6 | 3
Chills (General disorders) | 5 | 2
Pain (General disorders) | 7 | 0
Pyrexia (General disorders) | 6 | 0
Oedema peripheral (General disorders) | 3 | 0
Feeling jittery (General disorders) | 2 | 0
Malaise (General disorders) | 2 | 0
Asthenia (General disorders) | 1 | 0
Early satiety (General disorders) | 1 | 0
Feeling abnormal (General disorders) | 1 | 0
Gait disturbance (General disorders) | 1 | 0
Generalised oedema (General disorders) | 1 | 0
Injection site erythema (General disorders) | 0 | 1
Injection site haematoma (General disorders) | 1 | 0
Injection site irritation (General disorders) | 1 | 0
Injection site pruritus (General disorders) | 1 | 0
Injection site rash (General disorders) | 0 | 1
Local swelling (General disorders) | 1 | 0
Nodule (General disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 18 | 7
Pruritus (Skin and subcutaneous tissue disorders) | 21 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 7 | 2
Pruritus generalised (Skin and subcutaneous tissue disorders) | 5 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 0
Blister (Skin and subcutaneous tissue disorders) | 3 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 2 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 3 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 2 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 1
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Parakeratosis (Skin and subcutaneous tissue disorders) | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0
Scab (Skin and subcutaneous tissue disorders) | 0 | 1
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 28 | 7
Neutropenia (Blood and lymphatic system disorders) | 9 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 2
Lymphopenia (Blood and lymphatic system disorders) | 3 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 2 | 0
Pancytopenia (Blood and lymphatic system disorders) | 2 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Headache (Nervous system disorders) | 26 | 6
Dizziness (Nervous system disorders) | 12 | 2
Dysgeusia (Nervous system disorders) | 8 | 2
Syncope (Nervous system disorders) | 3 | 0
Hypersomnia (Nervous system disorders) | 1 | 1
Somnolence (Nervous system disorders) | 2 | 0
Tremor (Nervous system disorders) | 2 | 0
Amnesia (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 0
Disturbance in attention (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 1
Loss of consciousness (Nervous system disorders) | 1 | 0
Memory impairment (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 14 | 2
Irritability (Psychiatric disorders) | 9 | 2
Depression (Psychiatric disorders) | 9 | 1
Anxiety (Psychiatric disorders) | 3 | 3
Abnormal dreams (Psychiatric disorders) | 2 | 0
Mood swings (Psychiatric disorders) | 2 | 0
Anger (Psychiatric disorders) | 1 | 0
Libido decreased (Psychiatric disorders) | 1 | 0
Nightmare (Psychiatric disorders) | 0 | 1
Somnambulism (Psychiatric disorders) | 0 | 1
Stress (Psychiatric disorders) | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 9 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinitis atrophic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Blood creatinine increased (Investigations) | 7 | 1
Haemoglobin decreased (Investigations) | 3 | 2
Transaminases increased (Investigations) | 3 | 0
Weight increased (Investigations) | 2 | 1
Blood thyroid stimulating hormone decreased (Investigations) | 2 | 0
Blood triglycerides increased (Investigations) | 1 | 1
Blood urea increased (Investigations) | 2 | 0
Blood uric acid increased (Investigations) | 2 | 0
Platelet count decreased (Investigations) | 2 | 0
Weight decreased (Investigations) | 2 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Blood cholesterol increased (Investigations) | 0 | 1
Blood glucose decreased (Investigations) | 1 | 0
Blood glucose increased (Investigations) | 1 | 0
Blood potassium increased (Investigations) | 1 | 0
Blood pressure increased (Investigations) | 1 | 0
Glomerular filtration rate decreased (Investigations) | 0 | 1
Liver function test abnormal (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0
Serum ferritin decreased (Investigations) | 1 | 0
Skin turgor decreased (Investigations) | 1 | 0
Thyroxine increased (Investigations) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Sinusitis (Infections and infestations) | 4 | 1
Influenza (Infections and infestations) | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 1
Cellulitis (Infections and infestations) | 1 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 1
Nasopharyngitis (Infections and infestations) | 1 | 1
Oral candidiasis (Infections and infestations) | 2 | 0
Oral herpes (Infections and infestations) | 1 | 1
Pharyngitis (Infections and infestations) | 2 | 0
Rhinitis (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 2 | 0
Bronchitis (Infections and infestations) | 0 | 1
Furuncle (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Skin candida (Infections and infestations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 7 | 0
Gout (Metabolism and nutrition disorders) | 4 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 2 | 0
Increased appetite (Metabolism and nutrition disorders) | 2 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 2
Laceration (Injury, poisoning and procedural complications) | 2 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 2 | 0
Anal injury (Injury, poisoning and procedural complications) | 0 | 1
Bite (Injury, poisoning and procedural complications) | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Incision site rash (Injury, poisoning and procedural complications) | 1 | 0
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 | 1
Renal failure (Renal and urinary disorders) | 5 | 1
Urinary incontinence (Renal and urinary disorders) | 2 | 0
Bladder discomfort (Renal and urinary disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1
Vision blurred (Eye disorders) | 4 | 1
Orbital oedema (Eye disorders) | 1 | 0
Visual impairment (Eye disorders) | 1 | 0
Vitreous floaters (Eye disorders) | 1 | 0
Hypertension (Vascular disorders) | 3 | 2
Haematoma (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0
Palpitations (Cardiac disorders) | 2 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1
Autoimmune hepatitis (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 1 | 0
Ear discomfort (Ear and labyrinth disorders) | 1 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0
Cushingoid (Endocrine disorders) | 1 | 0
Liver transplant rejection (Immune system disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
It was decided by Sponsor on 13 January 2014 to terminate the study early at the primary efficacy endpoint (SVR12) as part of a decision to modify the drug development plan. Eligible participants completed virologic follow-up after termination.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI is free to publish results of the study after (1) the first multi-center publication, (2) if the sponsor elects not to publish the results, or (3) 18 months after close of the study, whichever occurs first. Proposed publications are to be submitted to the sponsor for review and comment for a period of at least 45 days (which may be extended under certain circumstances related to protection of intellectual property); the sponsor cannot require changes to the proposed publications.